CLINICAL TRIAL: NCT01734499
Title: The Change Cycle Intervention for Improving Quality of Life in Breast Cancer Survivors
Acronym: CCIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A12-3719
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Survivorship; Coping; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coping Class (Experimental): A 4-hour structured program which will be offered once a month as the "Coping Class" by a certified facilitator of "The Change Cycle." Quality of Life survey completed at 5 time points after informed consent.
  Interventions: Behavioral: Coping Class; Behavioral: FACT-B Quality of Life
- Standard of Care (Active Comparator): Standard of Care. Three components of this: (1)Surveillance Program, (2)Local support groups centered at community cancer centers, (3)Comprehensive Postoperative Rehabilitation which offers physical and occupational rehabilitation.Quality of Life surveys completed at 5 time points after informed consent.
  Interventions: Behavioral: Standard of Care; Behavioral: FACT-B Quality of Life

INTERVENTIONS:
Behavioral: Coping Class — A 4-hour structured program which will be offered once a month as the "Coping Class" by a certified facilitator of "The Change Cycle." The coping class uses standardized materials and skills training. Standardized materials for the intervention arm will include "Change Moves Me" Participant's Guide/Journal, Locator Assessment Profile, The Change Cycle Color Model, and class evaluation. The structure of the class includes a profile of each stage to gain perspective and understanding, teaching personal change skills for each stage and a primary focus for movement to the next stage. The overall design follows an "act as if" philosophy, guiding participants through each stage of The Change Cycle, irrespective of which stage they are actually in.
  Arms: Coping Class
Behavioral: Standard of Care — Standard of Care. Three components of this: (1)Surveillance Program: all patients diagnosed with breast cancer are seen every six months for the first two years and yearly thereafter to rule out disease recurrence by history and physical exam at each visit in addition to the annual mammogram. (2)Local support groups centered at community cancer centers. These are generally attended by 12-16 women monthly; all breast cancer patients receive the information about these groups. Associated with these programs, some classes are offered sporadically in nutrition, and exercise. (3)Comprehensive Postoperative Rehabilitation which offers physical and occupational rehabilitation to all women, thus provides prevention and treatment of lymphedema and monitored shoulder range of motion.
  Arms: Standard of Care
Behavioral: FACT-B Quality of Life — The FACT-B Quality of Life is a 44-item instrument that was developed by combining nine breast cancer-specific QL items with the FACT general QL instrument. The FACT-B consists of the following subscales: physical wellbeing (PWB), functional wellbeing (FWB), emotional wellbeing (EWB), social/family wellbeing (SWB), and breast cancer specific concerns (BCS).

SUMMARY:
This study is proposed to assess long-term Quality of Life issues in breast cancer survivors by measuring the impact on the quality of life made by the structured "Change Cycle Work Shop" coping class as compared to current local standard of care programs. It has been shown that breast cancer treatment can have long-term bio-psychosocial consequences. Specific evidence-based interventions are needed to address Quality of Life concerns in order to improve the overall outcome of breast cancer and its treatment beyond the focus on mortality rate.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among North American women. A combination of screening mammography and improvements in treatment has resulted in a substantial decrease in mortality which explains why more women diagnosed at a younger age are becoming long-term survivors.Consequently, quality of life (QL) issues have become increasingly important in the contemporary multidisciplinary management of breast cancer. Standard of car survivorship program has evolved over several years to include 3 facets: (1)clinical surveillance program to include routine follow up exams; (2) local support group programs; and (3) rehabilitation program offering physical and occupational rehab, along with lymphedema prevention and treatment.

Many studies have reported on successful interventions (listed in our references) with improvements in quality of life; however the effects did not last long after intervention. This has brought into question the real value of such interventions. The proposed class will focus on teaching life skills that have shown long-lasting effect in the corporate world of change. Thus, our goal is to determine if the impact of the class will be similar in the healthcare arena, specifically cancer survivorship. Our last study on assessing quality of life revealed that patients were suffering deficits in quality of life, specifically with regard to the emotional scale despite the standard of care approach available. We therefore propose this intervention to be studied as proof of concept so that depending on the results of the proposed trial, this class can become a routine part of the survivorship program.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 years old or older
* established diagnosis of breast cancer
* diagnosis from January 2010 onward
* must be patient of Texas Tech University Health Sciences Center-Breast Center of Excellence
* must agree to participate in study structure of randomization

Exclusion Criteria:

* those who do not accept randomization
* women with medical conditions that preclude them from attending the coping class
* women with personal issues that preclude them from attending the coping class

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | Baseline
Quality of Life Questionnaire | change from Baseline and at 6 months
Quality of Life Questionnaire | change from Baseline and at 12 months
Quality of Life Questionnaire | change from Baseline and at 18 months
Quality of Life Questionnaire | change from Baseline and at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rakhshanda L Rahman, MD, Principal Investigator — Texas Tech University Health Sciences Center-Amarillo
Locations (1):
- Texas Tech University Health Sciences Center, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Cancer Statistics Working Group. United States Cancer Statistics: 1999-2005 Incidence and Mortality Web-based Report. Atlanta (GA): Department of Health and Human Services, Centers for Disease Control and Prevention, and National Cancer Institute; 2009.http://www.cdc.gov/uscs.
- [Background] http://www.cancer.org/Research/CancerFactsFigures/CancerFactsFigures/cancer-facts-and-figures-2010 (accessed on 9/10/2011).
- [Background] http://statecancerprofiles.cancer.gov/prevalence/index.php?
- [Background] Garfinkel L, Boring CC, Heath CW Jr. Changing trends. An overview of breast cancer incidence and mortality. Cancer. 1994 Jul 1;74(1 Suppl):222-7. doi: 10.1002/cncr.2820741304. PMID 8004590
- [Background] De Angelis R, Tavilla A, Verdecchia A, Scoppa S, Hachey M, Feuer EJ, Mariotto AB. Breast cancer survivors in the United States: geographic variability and time trends, 2005-2015. Cancer. 2009 May 1;115(9):1954-66. doi: 10.1002/cncr.24217. PMID 19248047
- [Background] Brinton LA, Sherman ME, Carreon JD, Anderson WF. Recent trends in breast cancer among younger women in the United States. J Natl Cancer Inst. 2008 Nov 19;100(22):1643-8. doi: 10.1093/jnci/djn344. Epub 2008 Nov 11. PMID 19001605
- [Background] American Cancer Society. Cancer Facts and Figures 2009. American Cancer society: Atlanta, GA, 2009
- [Background] Meyerowitz BE. Psychosocial correlates of breast cancer and its treatments. Psychol Bull. 1980 Jan;87(1):108-31. No abstract available. PMID 7375595
- [Background] Glanz K, Lerman C. Psychosocial impact of breast cancer: A critical review. Ann Behav Med 14:204-212, 1992
- [Background] Bloom JR, Stewart SL, Chang S, Banks PJ. Then and now: quality of life of young breast cancer survivors. Psychooncology. 2004 Mar;13(3):147-60. doi: 10.1002/pon.794. PMID 15022150
- [Background] Ganz PA, Desmond KA, Leedham B, Rowland JH, Meyerowitz BE, Belin TR. Quality of life in long-term, disease-free survivors of breast cancer: a follow-up study. J Natl Cancer Inst. 2002 Jan 2;94(1):39-49. doi: 10.1093/jnci/94.1.39. PMID 11773281
- [Background] Borrelli B. The assessment, monitoring, and enhancement of treatment fidelity in public health clinical trials. J Public Health Dent. 2011 Winter;71 Suppl 1:S52-63. PMID 21656954
- [Background] Calman KC. Definitions and dimensions of quality of life. In Quality of life of cancer patients, Aaronson NK, Beckmann J (eds). Raven Press: New York, 1987; 1-10
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Stanton AL, Danoff-Burg S, Cameron CL, Bishop M, Collins CA, Kirk SB, Sworowski LA, Twillman R. Emotionally expressive coping predicts psychological and physical adjustment to breast cancer. J Consult Clin Psychol. 2000 Oct;68(5):875-82. PMID 11068973
- [Background] McCaul KD, Sandgren AK, King B, O'Donnell S, Branstetter A, Foreman G. Coping and adjustment to breast cancer. Psychooncology. 1999 May-Jun;8(3):230-6. doi: 10.1002/(SICI)1099-1611(199905/06)8:33.0.CO;2-#. PMID 10390735
- [Background] Schnoll RA, Harlow LL, Stolbach LL, Brandt U. A structural model of the relationships among stage of disease, age, coping, and psychological adjustment in women with breast cancer. Psychooncology. 1998 Mar-Apr;7(2):69-77. doi: 10.1002/(SICI)1099-1611(199803/04)7:23.0.CO;2-8. PMID 9589505
- [Background] Allen SM, Shah AC, Nezu AM, Nezu CM, Ciambrone D, Hogan J, Mor V. A problem-solving approach to stress reduction among younger women with breast carcinoma: a randomized controlled trial. Cancer. 2002 Jun 15;94(12):3089-100. doi: 10.1002/cncr.10586. PMID 12115339
- [Background] www.changecycle.com
- [Background] Kubler-Ross. On Death and Dying: What the Dying Have to Teach Doctors, Nurses, Clergy and their own Families. Simon and Schuster, New York, 1969
- [Background] Ellis A. MacLaren C. (1998). Rational-emotive behavior therapy: A therapist's guide. California: Impact publishers
- [Background] Piaget, J. and Inhelder, B. (1962). The Psychology of the Child. New York: Basic Books
- [Background] Argyris, C. (1994). Knowledge for Action. San Francisco CA: Jossey-Bass
- [Background] Apter, Michael J. Reversal theory: What is it? The Psycologist 1997; 10(5): 217-20
- [Background] Ellis A (1994). Reason and Emotion in psychotherapy-revised and updated. New York, NY: Birch Lane Press
- [Background] Schwartz, B. (2004). The paradox of choice: why more is less. New York: Ecco Press
- [Background] Iyengar SS, Lepper MR. When choice is demotivating: can one desire too much of a good thing? J Pers Soc Psychol. 2000 Dec;79(6):995-1006. doi: 10.1037//0022-3514.79.6.995. PMID 11138768
- [Background] Bridges W. (2003). Managing transitions: Making the most of change. 2nd ed. New York: Da Capo Press
- [Background] Collins J. (2001). Good to Great: Why some companies make the leap… and others don't. New York: Harper Business
- [Background] Maslow A. A theory of human motivation. Psychological Review 1943; (50(4): 370-96
- [Background] Trotter R. The Mystery of Mastery. Psychology Today 1986; 20(7): 32-8
- See also: United States Cancer Statistics: 1999-2005 Incidence and Mortality Web-based Report. — http://www.cdc.gov/uscs
- See also: Change Cycle — http://www.changecycle.com